CLINICAL TRIAL: NCT06595654
Title: Treatment of Negative Symptoms of Schizophrenia by Repetitive Transcranial Magnetic Stimulation: A Naturalistic Study
Brief Title: Treatment of Negative Symptoms of Schizophrenia by rTMS
Acronym: SN RENAT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre hospitalier de Ville-Evrard, France (Other)
Responsible Party: Principal Investigator, Dominique JANUEL, Head of clinical research unit, Centre hospitalier de Ville-Evrard, France
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2021-A02710-40
Record Dates: First submitted 2024-07-24; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Schizophrenia; Negative Symptoms in Schizophrenia
Keywords: rTMS; TMS; Transcranial magnetic stimulation; naturalistic
MeSH Terms: conditions — Schizophrenia | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Method 1 (Other): One stimulation session per day for 20 working days, so 4 weeks (frequency of 10 Hz, 80% 100% of motor threshold). Each session lasts 20 min. The duration of the train is 4 s, an inter-train of 56s.
  Interventions: Other: repetitive Transcranial Magnetic Stimulation
- Method 2 (Other): Two stimulations sessions per day, with 1 hour apart, for 20 working days, so 4 weeks (frequency of 20 Hz, 100% of motor threshold).Each session lasts 28 min. The duration of the train of 10 s, an inter-train of 80s The total number of pulses is 40000 in 20 trains or 2000 per day.
  Interventions: Other: repetitive Transcranial Magnetic Stimulation
- Method 3 (Other): Two stimulations session per day for 10 working days, so 2 weeks. The protocol is delivered in bursts containing 3 pulses at 50 Hz repeated at 200 ms intervals for 2 s (i.e., 5 Hz). Stimulation intensity is set at 80% of the idle motor threshold intensity
  Interventions: Other: repetitive Transcranial Magnetic Stimulation
- Method 4 (Other): Five to ten sessions per day, 50 minutes apart, with 90% SM for 10 working days, so 2 weeks. 1 of stimuli every 20 ms (50Hz) repeated 3 times, this train itself repeated every 200 ms (5 Hz) or 60 cycles of 10 blocks of 3 stimuli. The duration of the train is 2 seconds with an inter-train of 8 seconds. So there are 1800 stimuli per session
  Interventions: Other: repetitive Transcranial Magnetic Stimulation

INTERVENTIONS:
Other: repetitive Transcranial Magnetic Stimulation — * Patient is in a chair.
  * Hearing protection will be implemented.
  * The corresponding targeting method will be implemented.
  * The stimulation coil will be set up according to the indications of the targeting method.
  * A caregiver is present throughout the session.
  * After the session, the patient is re-assessed clinically for possible adverse effects.
  * If an adverse reaction is objectified, a doctor on site, is quickly mobilized.

SUMMARY:
The purpose of this study is to assess the effectiveness of rTMS on the negative symptoms of schizophrenia in real conditions. It will also provide a regulatory framework to rTMS treatments under these conditions. 4 types of rTMS protocols are proposed, allowing to adapt to patients and their tolerances.Treatment lasts between 2 and 4 weeks, with a follow-up period of 3 months after treatment to observe relapses.To assess the evolution of negative symptoms between baseline and the end of treatment, investigators use SANS (Scale for the Assessment of Negative Symptoms).

ELIGIBILITY:
Inclusion Criteria:

* Patient over 18 years of age
* Patient diagnosed with schizophrenia according to the DSM-V criteria (Diagnostic and Statistical Manual of Mental Disorder V5, 2013)
* Stable drug treatment for at least 4 weeks
* Presence or persistence of negative symptoms in the foreground:

Negative PANSS score ⩾21, positive PANSS score ⩽24

* Patient (or legal representative) willing to participate in the study and having signed an informed consent
* Patient fluent in the French language
* Affiliation to a social security scheme

Exclusion Criteria:

* Present a contraindication to TMS: intracranial foreign body, unstabilized epilepsy, cochlear implant, pace-maker
* Presence of an unstabilized medical condition
* Pregnant woman
* Woman of childbearing potential and without effective contraception
* Breastfeeding woman

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Estimated)
Dates: Start 2023-06-09 (Actual); Primary Completion 2027-09 (Estimated); Study Completion 2028-03 (Estimated)

PRIMARY OUTCOMES:
Evaluate the efectiveness of rTMS on the negative symptoms of schizophrena, assessed by the SANS ( Scale Assessment Negative Symptoms). | Baseline (day 1) to end of treatment (2 or 4 weeks)
  The SANS is a scale used for negative symptoms that is initially made up of 19 items divided into five sub-scales: emotional blunder, pedigree, avolition-apathy, anhedonia and social withdrawal. Based on the percentage reduction of this score after 2-4 weeks, patients will be allocated according to the following criteria:
  * Remission: 75%
  * Effective treatment: 50-74%
  * Improvement/response: 25-49%
  * No answer: <25%

SECONDARY OUTCOMES:
Evaluate the impact of this treatment on general psychopathology assessed by PANSS and CGI. | Baseline (day 1), end of treatment (2 or 4 weeks), 4 weeks, 12 weeks and 24 weeks after the end of treatment.
  The PANSS (Positive and Negative Syndrome Scale) is composed of 3 parts: positive symptoms, negative symptoms and general psychopathology. The last part consists of 16 items. The score can range from 16 to 112. The CGI (Clinical Global Impression) is a 3-item scale: the severity of the disease, the overall improvement and the efficiency index. The first two items are scored from 0 to 7, and the last in a 4x4 table.
Assess the impact of this treatment on response rate by the SANS | Baseline (day 1) to end of treatment (2 or 4 weeks)
  The Scale for the Assessment of Negative Symptoms (SANS) splits assessment into five domains (Affective flattening, Alogia, Avolition, Anhedonia, Attention). Within each domain it rates separate symptoms from 0 (absent) to 5 (severe). The response is defined by a 25-49% reduction in the initial score.
Assess the impact of this treatment on the rate of remission by the number of remission with the SANS | Baseline (day 1) to end of treatment (2 or 4 weeks)
  The Scale for the Assessment of Negative Symptoms (SANS) splits assessment into five domains (Affective flattening, Alogia, Avolition, Anhedonia, Attention). Within each domain it rates separate symptoms from 0 (absent) to 5 (severe). Based on the percentage reduction of this score after 2-4 weeks, patients will be considered in remission if they have a 75% reduction..
Assess the impact of this treatment on the relapse rate by the number of relapse with SANS | 4 weeks, 12 weeks and 24 weeks after the end of treatment.
  The SANS is a scale used for negative symptoms that is initially made up of 19 items divided into five sub-scales: emotional blunder, pedigree, avolition-apathy, anhedonia and social withdrawal. Based on the percentage reduction of this score after 2-4 weeks, patients will be allocated according to the following criteria:
  * Remission: 75%
  * Effective treatment: 50-74%
  * Improvement/response: 25-49%
  * No answer: <25%
Assess the impact of this treatment on cognitive symptoms by MOCA (Montreal Cognitive Assessment) and STROOP | Baseline (day 1) to end of treatment (2 or 4 weeks)
  The MoCA scale is the most sensitive rapid assessment test and provides the broadest evaluation of cognitive functions (attention, concentration, executive functions, memory, language, visualconstructive abilities, abstraction, calculation, orientation). A score < 26 (25 if cultural level < 3 = primary diploma = CEP) is considered abnormal.
  The Stroop scale evaluates the capacity for attention and inhibition; thus, it allows to measure the level of interference generated by the automatisms in the accomplishment of a task. The result of the test allows us to see if the person is correctly inhibiting the response (values greater than 0, positive) or if there are significant interference problems (if it is a negative value).
Assess the impact of this treatment on addictive attitudes by MCQ (Marijuana Craving Questionnaire) and CAST (Cannabis Abuse Screening Test) | Baseline (day 1) to end of treatment (2 or 4 weeks)
  The CAST is a 6-item scale for identifying problematic cannabis use. Each of these items describes use behaviors or problems encountered with cannabis use. The CAST score determines the patient's level of dependence. A score of 1 or less means low risk. A score of 2 means moderate risk. A score of 3 or higher means high risk. The MCQ self-report scale is a questionnaire on marijuana craving. It consists of four constructs or factors that characterize cannabis craving: compulsivity, emotionality, expectancy and determination. A separate score is calculated for each factor. The MCQ can be used to measure cue-induced craving in a research setting or natural craving in cannabis-dependent individuals presenting for treatment.
Assess the impact of this treatment on mood by CDSS (Calgary Depression Scale for Schizophrenia). | Baseline (day 1) to end of treatment (2 or 4 weeks)
  The CDSS, is designed to assess depression in people with schizophrenia. . The questionnaire consists of 9 items covering the last 2 weeks. Each item is evaluated on a 4 points Likert scale ranging from : "Absent" (0) to "Severe" (3). The total score is obtained by adding the items and gives a score out of 27.
Assess the impact of this treatment on quality of life by S-QoL-18 | Baseline (day 1), end of treatment (2 or 4 weeks), 4 weeks, 12 weeks and 24 weeks after the end of treatment.
  The SQoL questionnaire is a self-administered quality of life scale that assesses quality of life in people with schizophrenia from the patient's perspective. The questionnaire has 18 items, each item is rated on a 4 points Likert scale ranging from: "Much less" to "More than desired". Scores range from 0 to 100; higher scores represent better quality of life.
Assess the impact of this treatment on adverse reactions by the CGI | Baseline (day 1), end of treatment (2 or 4 weeks), 4 weeks, 12 weeks and 24 weeks after the end of treatment.
  The CGI (Clinical Global Impression) is a 3-item scale: the severity of the disease, the overall improvement and the efficiency index. The first two items are scored from 0 to 7, and the last in a 4x4 table. The last item allows a combined measurement of the main clinical effect and side effects.

CONTACTS AND LOCATIONS:
Overall Officials: Dominique Januel, Principal Investigator — Clinical research unit, EPS Ville Evrard
Locations (1):
- Etablissement Public de Santé de Ville-Evrard, Neuilly-sur-Marne, France

IPD SHARING:
Plan to Share IPD: No